CLINICAL TRIAL: NCT04040790
Title: Evaluation of Light Sensitivity and Visual Acuity Changes as Consequence of Rigid Gas Permeable (RGP) Scleral Contact Lenses With a Passive Artificial Iris
Brief Title: Performance of Rigid Gas Permeable (RGP) Scleral Contact Lenses With a Passive Artificial Iris
Acronym: RGPIRIS_PA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Several reasons: Financing ended before all study assessments were performed, covid-19 delayed design, production and shipment of IMD, experience gained during the study made it clear that lens design should be changed
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGPIRIS_PA
Record Dates: First submitted 2019-06-13; First posted 2019-08-01 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2021-11

CONDITIONS: Low Vision
Keywords: visual acuity; contrast sensitivity; scleral contact lens; artificial iris
MeSH Terms: conditions — Vision, Low | interventions — Tropicamide; Phenylephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Experimental): 15 healthy volunteers for trials with passive artificial iris
  Interventions: Device: Scleral contact lens without a passive artificial iris; Device: Scleral contact lens with a passive artificial iris with low contrast (<1:5); Device: Scleral contact lens with a passive artificial iris with high contrast (>1:5); Drug: Tropicamide and phenylephrine

INTERVENTIONS:
Device: Scleral contact lens without a passive artificial iris — Participants wear a scleral contact lens without a passive artificial iris (Design A) on the dominant eye to perform the baseline visual performance assessment
  Other Names: Control lens Design A
Device: Scleral contact lens with a passive artificial iris with low contrast (<1:5) — Participants wear a scleral contact lens with a low contrast (<1:5) passive artificial iris (Design B) on the dominant eye to perform the baseline visual performance assessment
  Other Names: Test lens Design B
Device: Scleral contact lens with a passive artificial iris with high contrast (>1:5) — Participants wear a scleral contact lens with a low contrast (<1:5) passive artificial iris (Design B) on the dominant eye to perform the baseline visual performance assessment
Drug: Tropicamide and phenylephrine — Participants receive pupil dilation eye drops on the dominant eye, after baseline measurement and before wearing the scleral contact lenses (Designs A, B and C)
  Other Names: Pupil dilation eye drops

SUMMARY:
Data from 15 healthy subjects will be recorded in two testing sessions spread on two days, using three lens designs (A, B and C). Before the measuring days, each subject will undergo an extra fitting session of a large-diameter scleral contact lens on the dominant eye, assessed by an experienced practitioner. The fitting data will be used to custom-make the three lens designs for each subject, thus ensuring their comfort and safety during the days of the experiments. During the experiment days baseline measurements will be obtained before and after pupil dilation and contact lens wear. During the first testing session data from the lens design A (reference lens without artificial iris) will be recorded. During the second testing session data from the lens designs B and C (lenses with artificial iris with different transmittances) will be recorded. In each testing session, contrast sensitivity and visual acuity will be evaluated and non-invasive imaging measurements will be undertaken (optical coherence tomography and slit lamp). A specific questionnaire will be given to the subject to assess comfort, light sensitivity, the horizontal visual angle and overall experience of the scleral lens and in combination with a pair of sunglasses category 3-4.

DETAILED DESCRIPTION:
First, the participant will be subjected to an RGP scleral contact lens fitting session, then during the second and third visits the participant will be subjected to several non-invasive procedures specific to the study in order to assess contrast sensitivity and visual acuity using the fitted and uniquely fabricated investigational medical devices. The tests will be performed after eye drops are supplied to dilate the pupil of the subjects (eye drops: tropicamide and phenylephrine). Besides the clinical experiments, the participant will be given a specific questionnaire in order to assess comfort, light sensitivity, horizontal visual angle and overall experience of the investigational medical device and in combination with a pair of sunglasses category 3-4. The investigators will document the occurrence of any adverse events and specific side effects during Day 2 and 3 (testing sessions with the investigational devices) in order to effectively assess their safety.

ELIGIBILITY:
Inclusion Criteria:

- Age between 18 and 45 years old

Exclusion Criteria:

* Iris disorders (i.e. ocular albinism, coloboma, aniridia).
* Known disease-related ocular surface problem (i.e. microbial keratitis).
* Known ocular pathologies (except refractive disorders).
* Coexistent ocular diseases impeding contact lens correction (i.e. glaucoma, previous ocular surgery).
* Corneal scarring.
* Low corneal endothelial cell count (< 1500 cells per mm2), with potential of corneal hypoxia-induced corneal edema induced by contact lens wear.
* Wearing of contact lenses in the last 24 hours (prior to the interventions).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Visual acuity assessment and comparison between Designs A, B and C by means of logMAR or equivalent value | 5 months from fitting session
  Compare visual acuity values obtained with different designs
Contrast sensitivity assessment and comparison between Designs A, B and C by means of threshold percentage or equivalent value | 5 months from fitting session
  Compare contrast sensitivity values obtained with different designs

SECONDARY OUTCOMES:
Device safety by comparing eventual adverse events with those found in scleral contact lenses | 5 months from fitting session
  Comparing adverse event of similar devices
Correct fitting | 5 months from fitting session
  Taking and analyzing ocular coherence tomography (OCT) images and slit lamp observations to estimate the clearance
Contact lens wear comfort, as assessed by subject data from questionnaires Rasch analyzed using a 4-Andrich ration scale model | 5 months from fitting session
  The subjective assessment will be carried out by means of questions on 3 content areas: lens comfort (3 questions), visual quality (4 questions) and general satisfaction with the lenses (3 questions).
Visual acuity assessment and comparison between Designs B (low contrast) and C (high contrast) by means of logMAR or equivalent value | 5 months from fitting session
  Comparing visual acuity between Designs B and C
Contrast sensitivity assessment and comparison between Designs B (low contrast) and C (high contrast) by means of threshold percentage or equivalent value | 5 months from fitting session
  Comparing contrast sensitivity between Designs B and C
Horizontal visual angle | 5 months from fitting session
  Angle at which the volunteer can see his fingers move when extending the arm (same side as dominant eye), 0°=arm extended to the side; 90°=arm straight ahead

CONTACTS AND LOCATIONS:
Overall Officials: Andres F Vasquez Quintero, Professor, Study Chair — University Ghent
Locations (1):
- University Hospital Ghent (UZGent), Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Lazaro S, Ferrer-Blasco T, Radhakrishnan H, Cervino A, Charman WN, Montes-Mico R. Visual function through 4 contact lens-based pinhole systems for presbyopia. J Cataract Refract Surg. 2012 May;38(5):858-65. doi: 10.1016/j.jcrs.2011.11.042. Epub 2012 Mar 16. PMID 22424803
- [Background] Pepose JS. Small-aperture contact lenses for presbyopia. J Cataract Refract Surg. 2012 Nov;38(11):2060-1; author reply 2062-4. doi: 10.1016/j.jcrs.2012.08.041. No abstract available. PMID 23079328
- [Background] Xu R, Gil D, Dibas M, Hare W, Bradley A. The Effect of Light Level and Small Pupils on Presbyopic Reading Performance. Invest Ophthalmol Vis Sci. 2016 Oct 1;57(13):5656-5664. doi: 10.1167/iovs.16-20008. PMID 27784070
- [Background] Eyeson-Annan ML, Hirst LW, Battistutta D, Green A. Comparative pupil dilation using phenylephrine alone or in combination with tropicamide. Ophthalmology. 1998 Apr;105(4):726-32. doi: 10.1016/S0161-6420(98)94030-1. PMID 9544648
- [Background] Compan V, Oliveira C, Aguilella-Arzo M, Molla S, Peixoto-de-Matos SC, Gonzalez-Meijome JM. Oxygen diffusion and edema with modern scleral rigid gas permeable contact lenses. Invest Ophthalmol Vis Sci. 2014 Sep 4;55(10):6421-9. doi: 10.1167/iovs.14-14038. PMID 25190661
- [Background] Holden BA, Mertz GW. Critical oxygen levels to avoid corneal edema for daily and extended wear contact lenses. Invest Ophthalmol Vis Sci. 1984 Oct;25(10):1161-7. PMID 6592160